CLINICAL TRIAL: NCT07089043
Title: A Single-Blind Dose-Ranging Study in Subjects With Neurogenic Orthostatic Hypotension to Evaluate the Effect of CST-3056 on Symptoms and Signs of Orthostatic Hypotension
Brief Title: A Study in Subjects With Neurogenic Orthostatic Hypotension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CuraSen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: CST3056-CLIN-021
Record Dates: First submitted 2025-07-14; First posted 2025-07-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Neurogenic Orthostatic Hypotension

STUDY DESIGN:
Intervention Model Description: This is a single-blind dose ranging study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CST-3056 (Experimental): Subjects will receive single doses of CST-3056 over 3 days and on the Optimal Dose Day (Day 5)
  Interventions: Drug: CST-3056
- Placebo (Placebo Comparator): Subjects will receive a single dose of placebo on 1 day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CST-3056 — Administered as an oral solution
  Arms: CST-3056
Drug: Placebo — Administered as an oral solution
  Arms: Placebo

SUMMARY:
This is a study to evaluate the effects of CST-3056 on orthostatic symptoms and signs in subjects with neurogenic orthostatic hypotension (nOH).

DETAILED DESCRIPTION:
This is a study to evaluate the effects of CST-3056 on orthostatic symptoms in subjects with nOH.

Subjects who use direct or indirect α1-AR agonists for treatment of nOH will need to discontinue those treatments for at least 1 day or 5 half-lives (whichever is longer) prior to assessment of orthostatic measures during Screening, and again prior to initiation of dosing for study drug on Day 1.

Following confirmation of eligibility, subjects will be enrolled and participate in a single-blind dose ranging study. Single oral doses of CST-3056 will be administered once-daily for five days (Days 1 through 4 and the Optimal Dose Day [Day 5]), as tolerated. The Individual Optimal Dose will be determined based on observations for each subject over Day 1 through Day 4, including standing blood pressure, and safety/tolerability of the dose.

Between 3-7 days after discharge from the in-patient stay, the Investigator or designee will contact the subject by telephone to review the subject's health status. Any adverse events reported by phone will be recorded and followed as medically appropriate as determined by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 and ≤ 85 years of age, at time of informed consent.
2. Diagnosed with symptomatic orthostatic hypotension due to Parkinson's disease or pure autonomic failure (i.e. neurogenic orthostatic hypotension).
3. At Screening, subjects must meet the diagnostic criteria of neurogenic orthostatic hypotension, as demonstrated by a decrease ≥20 mm Hg in systolic or ≥10 mm Hg in diastolic BP upon standing ≤3 minutes from a supine position.
4. At Screening, subjects must have a score ≥4 on the Orthostatic Hypotension Symptom Assessment (OHSA) scale question #1.
5. Currently receiving, or known to be responsive to, direct or indirect α1-AR agonists (e.g., midodrine, droxidopa) for treatment of nOH.
6. If the Investigator determines that additional autonomic function testing is required to confirm the diagnosis of autonomic dysfunction, the Valsalva maneuver may be performed to show the absence of BP overshoot during phase IV.
7. Body weight greater or equal to 50 kg and body mass index (BMI) between 18 and 35 kg/m2, inclusive at Screening.
8. Stable medical conditions for 3 months prior to Screening.
9. For patients taking antiparkinsonian medication: stable dose of levodopa, dopamine agonist, amantadine, and/or monoamine oxidase B inhibitor, i.e. unchanged for 1 month.
10. Subject is ambulatory with/without the use of an assistive device.
11. Willing to follow the protocol requirements and comply with protocol restrictions.
12. Capable of providing informed consent and complying with study procedures.
13. Able to speak, understand, and read English.

Exclusion Criteria:

1. Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathy of unknown significance, and autoimmune neuropathies.
2. Concomitant use of vasoconstricting agents for the purpose of increasing blood pressure (BP) such as ephedrine, dihydroergotamine, or midodrine must be stopped at least 1 day or 5 half-lives (whichever is longer) prior to dosing on Day 1 and throughout the duration of the study. Fludrocortisone use in the study will be limited to a stable dose of 0.1 mg once-daily (QD).
3. Supine SBP ≥ 170 mm Hg or seated SBP ≥ 140 mm Hg at Screening.
4. Subjects with clinically meaningful urinary retention who use or are likely to use α1-AR antagonists (e.g., tamsulosin [Flomax]), or other medications (e.g., trazodone).
5. Concomitant use of anti-hypertensive medication for the treatment of essential hypertension unrelated to autonomic dysfunction.
6. Evidence of any significant or unstable clinical disorder or laboratory finding that renders the subject unsuitable for receiving an investigational drug including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine (excluding managed hypo and hyperthyroidism), metabolic, renal, or other systemic disease or laboratory abnormality.
7. History of malignant disease within 5 years, including solid tumors and hematologic malignancies (except [a] basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured; [b] low-grade adenocarcinoma of the prostate).
8. Any clinically significant illness or disease (apart from those typically associated with neurodegenerative disease) as determined by medical and surgical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory assessments conducted at Screening.
9. History of suicidal ideation or an episode of clinically severe depression as determined by the Investigator.
10. Clinically significant abnormalities of ECG, including QTcF > 450 ms, for males and QTcF > 470 ms for females, and/or HR < 50 beats per minute, or evidence of clinically significant bundle branch blocks, as indicated by 12-lead ECG in a supine position at Screening.
11. A calculated eGFR of ≤60 mL/min/1.73m2 according to the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) equation at Screening.
12. Current use of any prohibited prescription medication during Screening or throughout study, unless approved by both the Investigator and the Sponsor Medical Monitor.
13. Prior treatment with any investigational drug ≤90 days prior to dosing (Day 1), or ≤5 half-lives of the drug (whichever is longer), or current enrollment in any other study treatment or disease study, except for observational studies.
14. Known or suspected alcohol or substance abuse within the past 12 months and/or positive test for alcohol or drugs of abuse at Screening.
15. Positive screening test for human immunodeficiency virus (HIV), hepatitis C antibody (HCV Ab) or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HbsAg] at Screening).
16. Females who are breastfeeding.
17. Any other reason for which the Investigator considers it is not in the best interest of the subject to undertake the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Standing Systolic Blood Pressure | Baseline and 1, 2, 3, and 4 hours post-dose on Days 1 to 4
  Baseline is defined as the pre-dose measurement on Day 1

SECONDARY OUTCOMES:
Change from Baseline in Seated Systolic Blood Pressure relative to placebo | Baseline and 5 minutes post-dose on Days 1 to 4
  Baseline is defined as the pre-dose measurement on Day 1
Change from Baseline in the Orthostatic Hypotension Symptom Assessment (OHSA) Question #1 relative to placebo | Baseline and 3 hours post-dose on Days 1 to 4
  The question asks subjects to rate the severity of their orthostatic hypotension symptoms (dizziness, lightheaded, feeling faint, or felling like you might black out) on an 11-point scale from 0-10, with 0 indicating no symptoms/no interference and 10 indicating the worst possible symptoms/complete interference. A higher score indicates a worse outcome. Baseline is defined as the pre-dose measurement on Day 1.
Change from Baseline in the heads-up tilt table test (HUTT) | Baseline and 3 hours post-dose on Optimal Dose Day (Day 5)
  Subjects will have blood pressure and heart rate measured continuously and/or intermittently after resting in the supine position and pre-dose measurements will be taken twice. After dosing, subjects will undergo a graded HUTT at 30, 45 and 60 degrees. Measurements will be taken continuously and/or intermittently and at 1 and 3 minutes after each degree of tilt.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — CuraSen Therapeutics, Inc.
Locations (3):
- United States (3):
  - CuraSen Investigational Site, Eatontown, New Jersey
  - CuraSen Investigational Site, New York, New York
  - CuraSen Investigational Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No